CLINICAL TRIAL: NCT07201077
Title: Overcoming Instrumentation Challenges in Real-World Uniportal Video-Assisted Thoracoscopic Surgery: A Prospective, Randomized, Controlled Trial Evaluating the SurgeoFlex Grasp Versus the Traditional Endograsper for Systemic Lymph Node Dissection in Patients With Early-Stage Non-Small Cell Lung Cancer
Brief Title: ArticuGrasp Trial: New Flexible Tool vs Standard Grasper for Lung Cancer Node Removal in Keyhole Chest Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jianxing He (Other)
Responsible Party: Sponsor-Investigator, Jianxing He, Professor and Chair, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ES-2025-165-01
Record Dates: First submitted 2025-08-15; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: SurgeoFlex grasp; Systematic lymph node dissection; Uniportal video-assisted thoracoscopic surgery; Minimally invasive thoracic surgery; Lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SurgeoFlex Grasp (SFG) (Experimental): Participants receive UVATS with SurgeoFlex Grasp for lymph-node dissection.
  Interventions: Device: Articulating lymph-node grasper (SurgeoFlex Grasp)
- Traditional Endograsper (TER) (Active Comparator): Participants receive UVATS with Traditional Endograsper for lymph-node dissection.
  Interventions: Device: Arm 2 Intervention Name Traditional rigid endograsper

INTERVENTIONS:
Device: Articulating lymph-node grasper (SurgeoFlex Grasp) — Arm 1 - SurgeoFlex Grasp A single-use, low-profile articulating grasper with a 5-millimetre (mm) shaft and a 360-degree (360°) steerable distal tip. During uniportal video-assisted thoracoscopic surgery (UVATS), the device is introduced through the same 3-4-centimetre (cm) utility incision used for the camera and stapler. The flexible neck allows the jaws to approach hilar and mediastinal lymph nodes from multiple angles without repositioning the instrument shaft, thereby reducing instrument collision and chest-wall torque.
  Arms: SurgeoFlex Grasp (SFG)
Device: Arm 2 Intervention Name Traditional rigid endograsper — Arm 2 - Traditional Rigid EndoGrasper A reusable, straight-shafted 5 mm grasper with fixed-angle jaws identical to those used in conventional multi-port video-assisted thoracoscopic surgery (VATS). The instrument is passed through the single 3-4 cm incision in the same fashion as the SurgeoFlex Grasp, but its rigid shaft limits the working angle and often requires external repositioning of the entire instrument to reach deep lymph-node stations.
  Arms: Traditional Endograsper (TER)

SUMMARY:
This study is testing whether a new, flexible surgical tool-the SurgeoFlex Grasp-makes keyhole chest operations for early-stage lung cancer easier, faster, and safer than the standard rigid tool used today.

What is the problem? In keyhole (uniportal) chest surgery, formally known as single-port video-assisted thoracoscopic surgery (VATS), surgeons reach the lung through one small incision between the ribs. Because the operating space is tight, the usual stiff instruments can bump into each other and into surrounding tissues. This difficulty can prolong lymph-node removal and increase the risk of complications.

What is being tested?

The trial compares two handheld tools:

SurgeoFlex Grasp (intervention): a slim, bendable grasper that can be steered around corners.

Traditional EndoGrasper (control): a straight, rigid grasper currently used as the standard.

Who is taking part? Approximately 100 adults with early-stage non-small-cell lung cancer (NSCLC) (tumours 3 cm or smaller) who are scheduled for keyhole surgery at The First Affiliated Hospital of Guangzhou Medical University.

What will happen?

Participants are allocated by randomisation into one of two groups:

SurgeoFlex group-surgeons use the new flexible tool. Control group-surgeons use the standard rigid tool. All other aspects of the operation, anaesthesia, and post-operative care remain identical for both groups.

What is measured? Lymphadenectomy time (duration required to remove the specified lymph nodes). Number of lymph nodes successfully removed. Frequency of surgical-instrument collisions or interference (instrument-clash events).

Surgeon workload during the operation (assessed with the National Aeronautics and Space Administration Task Load Index [NASA-TLX]).

Skin-incision length, pain scores (Visual Analogue Scale [VAS]), recovery time, infection rates, and overall cost.

Quality-of-life scores one month after surgery (European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaire Core 30 [EORTC QLQ-C30] and its lung-cancer module [EORTC QLQ-LC13]).

What is expected? The investigators expect the SurgeoFlex Grasp to shorten operative time, reduce instrument interference, lower surgeon stress, and accelerate recovery without increasing cost.

How will this help patients? If the new tool performs as anticipated, future patients undergoing keyhole lung-cancer surgery may experience shorter operations, smaller scars, less pain, and lower infection risk while still obtaining complete cancer-related lymph-node removal.

Where is the study taking place? The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, China.

Contact for more information:

Clinical Research Management Committee 151 Yanjiang Road, Yuexiu District, Guangzhou 510120, China Email: crmc@gzhmu.edu.cn

ELIGIBILITY:
Eligibility Criteria

Inclusion Criteria

* Age 18-70 years, any sex
* BMI 18.5-30 kg/m²
* Newly diagnosed non-small-cell lung cancer with pre-operative clinical stage cT1-2N0-1M0
* Scheduled to undergo single-port video-assisted thoracoscopic lobectomy with systematic lymph-node dissection
* Major organ function sufficient for surgery
* Written informed consent provided

Exclusion Criteria

* Small-cell lung cancer or mixed-type lung cancer
* Tumor invasion of main bronchus, chest wall, diaphragm, or major mediastinal vessels
* Previous ipsilateral thoracic surgery or prior neoadjuvant chemotherapy, radiotherapy, targeted therapy, or immunotherapy
* Severe cardiopulmonary dysfunction (FEV₁ <50 % predicted or LVEF <40 %)
* Pregnant or breastfeeding women
* Participation in another interventional clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Duration of Systemic Lymph Node Dissection (SLND) | Intraoperative; measured from the start of the first lymph node packet dissection to the completion of the final packet removal, up to a maximum of 60 minutes.

SECONDARY OUTCOMES:
Number of Lymph Nodes Retrieved | Intraoperatively, assessed immediately after the completion of systemic lymph node dissection.
Instrument Collision Counts | Intraoperatively, continuously recorded during systemic lymph node dissection and averaged per case.
Surgeon Cognitive Load (NASA-TLX score) | Intra-operatively, within 10 minutes after skin closure.
  National Aeronautics and Space Administration Task Load Index (NASA-TLX). The NASA-TLX is a multidimensional assessment tool that rates perceived workload across six subscales to assess a task's mental, physical, and temporal demands, as well as the performer's effort, frustration, and performance. The subscale ratings are combined into a weighted composite score. Range: 0-100 points (weighted composite of 6 subscales). Interpretation: Higher scores indicate greater perceived workload.
Skin Incision Length | At the end of the operation, before skin closure.
Post-operative Pain Score (0-10 numeric rating scale) | Daily during the first 3 post-operative days.
Incidence of Post-operative Infections | Within 30 days after surgery.
Operating Room Occupancy Time | Time Frame: Intra-operatively, from skin incision to wound closure, up to 6 hours.
Health-related Quality of Life (SF-36 score) | Assessed 1 month after surgery.
  36-Item Short-Form Health Survey (SF-36) quality-of-life score. The SF-36 is a standardized, self-administered survey evaluating eight health domains: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. Range: 0-100 points (each of the 8 domains is scored 0-100). Interpretation: A higher score indicates a better health status and quality of life.
Incidence of Device Malfunction | From device insertion to device removal, assessed continuously during each operation.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No